CLINICAL TRIAL: NCT02980003
Title: PrevenTion of Contrast-inducEd nephroAThy With urinE Alkalinization: the TEATE Study
Brief Title: PrevenTion of Contrast-inducEd nephroAThy With urinE Alkalinization
Acronym: TEATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Raffaele De Caterina, Principal Investigator, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TEATE study
Record Dates: First submitted 2016-11-05; First posted 2016-12-02 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Acute Kidney Injury; Contrast Media Reaction
Keywords: contrast media; contrast-induced acute kidney injury (AKI); contrast-induced nephropathy (CIN)
MeSH Terms: conditions — Acute Kidney Injury | interventions — Sodium Chloride; Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- isotonic saline (Active Comparator): patients will start hydration with isotonic saline 6 hours before angiography and continue for 12 hours after the procedure. The infusion rate will be 1 mL/kg/h in the first 5 hours they will receive isotonic saline at 1 mL/kg/h (reduced to 0.5 mL/kg/h if with ejection fraction <35% or New York Heart Association (NYHA) functional class III or IV). Then, will be infused at 3 mL/kg/h for 1 hour immediately before contrast medium injection; following this, patients will receive the same fluid at a rate of 1 mL/kg/h
  Interventions: Drug: isotonic saline
- i.v. sodium bicarbonate (Active Comparator): in the first 5 hours patients will receive isotonic saline at 1 mL/kg/h (reduced to 0.5 mL/kg/h if with ejection fraction <35% or NYHA functional class III or IV). Then, a solution of 1.4% sodium bicarbonate (167 mEq/L; 334 milliosmol (mOsm/L)) will be infused: the initial intravenous bolus will be 3 mL/kg/h for 1 hour immediately before contrast medium injection; following this, patients will receive the same fluid at a rate of 1 mL/kg/h (reduced to 0.5 mL/kg/h if with ejection fraction <35% or NYHA functional class III or IV) during the exposure to contrast and for 6 hours after the procedure. Later, patients will resume hydration with isotonic saline for further 6 hours.
  Interventions: Drug: i.v. sodium bicarbonate
- oral sodium bicarbonate: (Experimental): patients will start hydration with isotonic saline as well as Arm Hydration Alone. One hour before the angiography and 3 hours after patients will receive oral sodium bicarbonate at the dose of 4 g (47.6 mEq) dissolved in 60 mL of water. The drug will be weighed with a precision balance with a sensitivity of ± 0.1 mg and placed in a labeled sterile plastic container. The label will report the lot number, expiry date of the sodium bicarbonate lot, the signature of the pharmacist carrying out the weighing process, a serial number to identify the sample and the patient identification number.
  Documentation will be stored in the Laboratory of Galenic Preparations, Pharmacy Division, of the hospital.
  Interventions: Drug: oral sodium bicarbonate

INTERVENTIONS:
Drug: isotonic saline — patients will start hydration with isotonic saline 6 hours before angiography and continue for 12 hours after the procedure.
  Other Names: Isotonic sodium chloride solution
  Arms: isotonic saline
Drug: i.v. sodium bicarbonate — patients will start hydration with isotonic saline 6 hours before angiography and continue for 12 hours after the procedure. The patient receives solution of 1.4% sodium bicarbonate (167 mEq/L; 334 mOsm/L) one hours and six hours after procedure.
  Other Names: HCO3
  Arms: i.v. sodium bicarbonate
Drug: oral sodium bicarbonate — patients will start hydration with isotonic saline 6 hours before angiography and continue for 12 hours after the procedure. One hour before the angiography and 3 hours after patients will receive oral sodium bicarbonate at the dose of 4 g (47.6 mEq) dissolved in 60 mL of water
  Other Names: HCO3
  Arms: oral sodium bicarbonate:

SUMMARY:
Intravascular administration of iodinated contrast media is an essential tool for cardiovascular imaging and percutaneous coronary interventions. Nonetheless, the increasing incidence of contrast-induced nephropathy (CIN) has become an important and prognostically relevant problem along with the spreading of diagnostic and interventional procedures. CIN is largely dependent on oxidative damage and represents a considerable cause of renal failure, being associated with prolonged hospitalization and significant morbidity/mortality. The most effective treatment strategy of this serious complication remains prevention, and several preventive measures have been extensively investigated in the last few years. Pre-procedural hydration is the best known and mostly accepted strategy. The administration of sodium bicarbonate (HCO3) has controversial effects, and is likely to be ineffective when the infused dose is unable to achieve adequate urine alkalinization. Since alkaline pH suppresses the production of free radicals, increasing urine pH would be an attractive goal for CIN prevention. In a randomized clinical trial the investigators will test the hypothesis that urine alkalinization with either oral or i.v. bicarbonate on top of hydration alone is the main determinant of CIN prevention in a population of patients with moderate or severe chronic kidney disease scheduled for coronary angiography and/or angioplasty. If the investigators, demonstrate non-significant differences in urine alkalinization (primary endpoint) and incidence of CIN (secondary endpoint) between the bicarbonate groups, a practical implication will be that oral administration is preferable for practical reasons over the administration of i.v. bicarbonate.

DETAILED DESCRIPTION:
Contrast medium-induced nephropathy (CIN) is a recognized complication in coronary diagnostic and interventional procedures, and is associated with prolonged hospitalization and adverse clinical outcomes. The frequency of CIN ranges from 2% in low-risk patients to 50% in high-risk patients. The most important risk factors for CIN development are pre-existing renal failure, diabetes, age, volume and type of contrast medium. There are two main pathogenetic mechanisms postulated to cause CIN:

1. a direct toxic action of contrast medium on kidney tubule cells, causing a disruption of mitochondrial function, the generation of reactive oxygen species, and subsequent cell injury and apoptosis;
2. vasoconstriction, reducing the blood flow through the renal medulla and causing ischemia with cell damage The treatment of CIN is exclusively supportive. Treatment is particularly recommended in patients with chronic kidney disease (CKD - mild, moderate or severe, according to estimated glomerular filtration rate - eGFR). Several approaches have been tested in the prevention of CIN with variable success. Adequate hydration is widely accepted as the best method for prevention of CIN, and is today the only strategy generally accepted by international guidelines (class of recommendation I, level of evidence A). The use of N-acetyl cysteine, recommended even in the recent past, is not supported by a recent randomized trial14 and a meta-analysis. Hemodialysis and hemofiltration may be effective in preventive CIN, but are reserved to high-risk patients. Attempts at preventing CIN with various medications, such as furosemide, vitamin C, statins and numerous other, have been largely unsuccessful. The efficacy of bicarbonate in the prevention of CIN has been extensively tested; the rationale is here that urine alkalinization suppresses the formation of free radicals. Actually, studies on bicarbonate have been controversial, varying from beneficial to toxic effects; this could bring into question the role of alkalinizing procedures in preventing CIN. Nevertheless, favorable results of prevention protocols using bicarbonate have been noted in studies also documenting a significant alkalinization of urines; while a similar protocol did not prove to be effective when the dose of bicarbonate was insufficient to such aim. Moreover, Markota et al., in a recent study on patients with estimated eGFR >15 mL/min/1.73 m2 and scheduled for coronary angiography, after documenting that Na/K citrate significantly reduced the incidence of CIN when compared with hydration alone, have shown that patients having a urine pH <6 had a more than ten-fold higher incidence of CIN compared with patients whose urine pH was >6.28 These results confirm the potential role of urine alkalinization in preventing CIN and place the oral administration of alkalinizing drugs as an attractive method compared to the more complex, and not always effective, i.v. infusion of bicarbonate. Finally, oral doses of bicarbonate may be sufficient to alkalinize the urine and thus to prevent CIN. In a study recently published, an oral dose of 4 g was sufficient to obtain, two hours after administration, an adequate urinary alkalinization with a pH >7 in all participants without side effects. This value was maintained and even magnified nearly 8 hours after the last dose. Interestingly, the Authors observed an additive effect after the second dose, showing a nondepleting urine pH, despite the reported short half-life of sodium bicarbonate.

Against this background, the investigators will here test the hypothesis that both oral and i.v. bicarbonate are adequate strategies for CIN prevention in patients after coronary angiography. Comparing the incidence of CIN according to urine pH achieved immediately before angiography, the investigators aim at demonstrating that urine alkalinization is the real goal, and that results are here largely independent from the strategy adopted to achieve it. The investigators will therefore compare the efficacy in alkalinizing urine and preventing CIN of three different strategies: hydration alone; hydration plus i.v. sodium bicarbonate; and hydration plus oral bicarbonate. Favorable results of the bicarbonate groups compared to the control group could increase the evidence supporting the use of alkalinizing strategies to prevent CIN; at the same time, non-inferiority results of the oral group compared to i.v. bicarbonate group could suggest the more practical oral administration as the preferred prevention strategy.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients scheduled for coronary angiography and/or angioplasty;
* eGFR <60 mL/min/1.73 m2, but >15 mL/min/1.73 m2 (MDRD formula).

Exclusion Criteria:

* acute renal insufficiency;
* emergency catheterization (e.g., STEMI patients) preventing the possibility of pretreatments;
* a history of adverse reactions to contrast media;
* use of potentially nephrotoxic drugs (non-steroidal anti-inflammatory drugs, aminoglycosides, sulphonamides, cyclosporin, tacrolimus, methotrexate or platinum complexes) from 48 hours before to 24 hours after the procedure, but allowing drugs deemed essential for cardiovascular therapy (diuretics, acetylsalicylic acid, angiotensinconverting enzyme inhibitors, angiotensin receptor blockers or aliskiren);
* pulmonary edema;
* multiple myeloma and other monoclonal gammopathies;
* factors predisposing to kidney injury: diarrhea, vomiting, dehydration or bleeding;
* exposure to contrast media within 7 days before the procedure; pregnancy; -
* hypersensitivity to the active substance or to any of the excipients;
* Metabolic or respiratory alkalosis, particularly if hypochloremic (vomiting, gastrointestinal losses, diuretic therapy);
* Hypocalcemia;
* use of N-acetyl cysteine, theophylline, dopamine, fenoldopam, mannitol, citrate or bicarbonate within 48 hours before coronary angiography;
* Chronic and / or acute therapy with corticosteroid, quinidine, ephedrine and pseudoephedrine;
* urinary tract infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-03; Primary Completion 2020-10-30 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
The incidence of CIN according to urine alkalinization achieved immediately before angiography | 48 hours after randomization
  The investigators primary hypothesis is that the incidence of CIN definition is significantly different in patients achieving urine alkalinization compared with patients not achieving it.

SECONDARY OUTCOMES:
Urine PH | 48 hours after randomization
  The investigators hypothesis is that the proportion of patients achieving urine alkalinization (pH >6) will be greater in patients allocated to the sodium bicarbonate group or the oral sodium/potassium citrate group compared to the control group
the incidence of CIN in three treatment groups | 48 hours after coronary angiography
  The investigators hypothesis is that the proportion of patients that develop a CIN will be greater in patients allocated to the control group compared to patients assigned to other groups
non-inferiority comparison between oral sodium bicarbonate group and i.v. sodium | 48 hours after coronary angiography
  The non-inferiority of oral bicarbonate group respect to i.v. sodium bicarbonate group will be evaluated in term of incidence of CIN.
non-inferiority comparison between oral sodium bicarbonate group and i.v. sodium bicarbonate | 48 hours after coronary angiography
  the non-inferiority of oral bicarbonate group respect to i.v. sodium bicarbonate group will be evaluated in term of proportion of patients achieving urine alkalinization

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele De Caterina, Principal Investigator — G. d'Annunzio University
Locations (1):
- Institute of Cardiology - Center of Excellence on Aging, G. d'Annunzio University, Chieti, CH, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Parfrey PS, Griffiths SM, Barrett BJ, Paul MD, Genge M, Withers J, Farid N, McManamon PJ. Contrast material-induced renal failure in patients with diabetes mellitus, renal insufficiency, or both. A prospective controlled study. N Engl J Med. 1989 Jan 19;320(3):143-9. doi: 10.1056/NEJM198901193200303. PMID 2643041
- [Result] Merten GJ, Burgess WP, Gray LV, Holleman JH, Roush TS, Kowalchuk GJ, Bersin RM, Van Moore A, Simonton CA 3rd, Rittase RA, Norton HJ, Kennedy TP. Prevention of contrast-induced nephropathy with sodium bicarbonate: a randomized controlled trial. JAMA. 2004 May 19;291(19):2328-34. doi: 10.1001/jama.291.19.2328. PMID 15150204
- [Result] Markota D, Markota I, Starcevic B, Tomic M, Prskalo Z, Brizic I. Prevention of contrast-induced nephropathy with Na/K citrate. Eur Heart J. 2013 Aug;34(30):2362-7. doi: 10.1093/eurheartj/eht009. Epub 2013 Jan 24. PMID 23349296
- [Result] Rihal CS, Textor SC, Grill DE, Berger PB, Ting HH, Best PJ, Singh M, Bell MR, Barsness GW, Mathew V, Garratt KN, Holmes DR Jr. Incidence and prognostic importance of acute renal failure after percutaneous coronary intervention. Circulation. 2002 May 14;105(19):2259-64. doi: 10.1161/01.cir.0000016043.87291.33. PMID 12010907
- [Derived] Lombardi M, Molisana M, Genovesi E, De Innocentiis C, Limbruno U, Misuraca L, Moretti L, Di Vito L, Renda G, Zimarino M, Di Nicola M, De Caterina R. Urine alkalinisation to prevent contrast-induced acute kidney injury: the prospective, randomised, controlled, open-label TEATE trial. EuroIntervention. 2022 Sep 20;18(7):562-573. doi: 10.4244/EIJ-D-22-00010. PMID 35620986